CLINICAL TRIAL: NCT06028451
Title: ManagemEnt of Antifungal Drug in Invasive Aspergillosis：a Real-word Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Other Study IDs: 2023ZDSYLL357-P01
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Invasive Aspergillosis
Keywords: invasive aspergillus infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Critically ill patients with invasive aspergillus infection who survived
  Interventions: Other: Record the information data
- Nonsurvivors: Critically ill patients with invasive aspergillus infection who not survived
  Interventions: Other: Record the information data

INTERVENTIONS:
Other: Record the information data — Record the information data

SUMMARY:
To assessed the current situation and outcome of critically ill patients with invasive aspergillus infection.

DETAILED DESCRIPTION:
To assessed the current situation and outcome of critically ill patients with invasive aspergillus infection.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 year-old
* Diagosed as invasive aspergillus infection

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagosed as invasive aspergillosis
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 day

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Southeast University
Locations (1):
- Southeast University, Zhongda hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided